CLINICAL TRIAL: NCT02095171
Title: A Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Study of PRX002 Administered by Intravenous Infusion in Healthy Subjects
Brief Title: Single Ascending Dose Study of PRX002 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Prothena Biosciences Limited (Industry)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRX002-CL001
Record Dates: First submitted 2014-03-14; First posted 2014-03-24 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-02

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- PRX002 (Experimental)
  Interventions: Drug: PRX002
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: PRX002
  Arms: PRX002
Other: Placebo
  Arms: Placebo

SUMMARY:
This single ascending dose study is to determine safety, tolerability, pharmacokinetics and immunogenicity of PRX002 in approximately 40 healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects
* Body mass index (BMI) between 18-32 kg/m2 with a minimum weight of 46 kg
* Female subjects must be surgically sterile or post-menopausal or if of child-bearing potential must use contraception
* Male subjects and their partners of childbearing potential must use contraception

Exclusion Criteria:

* Positive test for drug of abuse
* Past or current history of alcohol abuse
* Positive for hepatitis B, hepatitis C or HIV infection

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-03; Primary Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability as determined by number of subjects with adverse events | up to 3 months
Determination of pharmacokinetics parameters | up to 3 months
  - maximum concentration (Cmax)
Determination of pharmacokinetics parameters | up to 3 months
  - time of the maximum measured concentration (Tmax)
Determination of pharmacokinetics parameters | up to 3 months
  - area under the concentration-time curve from time zero to the last quantifiable concentration time-point (AUClast)
Determination of pharmacokinetics parameters | up to 3 months
  - area under the concentration-time curve from time zero extrapolated to infinity (AUCinf)
Determination of pharmacokinetics parameters | up to 3 months
  - elimination rate constant
Determination of pharmacokinetics parameters | up to 3 months
  - terminal elimination half life (t½)
Determination of pharmacokinetics parameters | up to 3 months
  - clearance (CL)
Determination of pharmacokinetics parameters | up to 3 months
  - apparent volume of distribution (Vd)

SECONDARY OUTCOMES:
Immunogenicity as determined by measurement of anti-PRX002 antibodies | up to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Neumann, PhD, Study Director — Clinical Trials Prothena Biosciences Inc
Locations (1):
- San Antonio, Texas, United States